CLINICAL TRIAL: NCT07223463
Title: A Tailored Medication Adherence-Promotion Intervention for Adolescents and Young Adults With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Seattle Children's Hospital (Other); University of Kansas Medical Center (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R37CA302422 (NIH); R37CA302422 (NIH)
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Medication Adherence
Keywords: adolescents and young adults; cancer; adherence
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Program (Experimental): 8-week program including 4 coach visits and 4 text check-ins
  Interventions: Behavioral: Tailored Program
- Feedback Program (Uniform Standard of Care) (Other): 8-week feedback program including weekly texts
  Interventions: Behavioral: Feedback Program (Uniform Standard of Care)

INTERVENTIONS:
Behavioral: Tailored Program — Participants will participate in 4 sessions with a coach, 1 every other week. During these sessions, the participant will work with their coach to identify a barrier to adherence they would like to target. Then, they will work with their coach to create an action plan using evidence-based behavior change techniques to address this barrier. In between sessions (on alternating weeks), the coach will check-in with a text reminder about the plan.
  Arms: Tailored Program
Behavioral: Feedback Program (Uniform Standard of Care) — Participants will receive weekly text messages with feedback about their adherence and guidance for requesting additional support if desired
  Arms: Feedback Program (Uniform Standard of Care)

SUMMARY:
The goal of this clinical trial is to learn if a tailored intervention can help make it easier for adolescents and young adults with cancer to take their medications. The main questions the researchers are trying to answer are:

* Does the tailored intervention increase adherence?
* Does the tailored intervention improve quality of life?
* Does the tailored intervention reduce health care utilization?

The researchers will compare the tailored intervention to a uniform standard of care intervention (an intervention designed to be similar to what is currently happening in clinical care) to see if the tailored intervention works to improve adherence.

Participants will:

* Use an electronic pill bottle or box to store their medication
* Participate in intervention sessions
* Complete surveys before the intervention, after the intervention, and 6-months later

DETAILED DESCRIPTION:
The proposed research includes a randomized clinical trial of a tailored adherence-promotion intervention (Tailored Program) as compared to uniform standard of care (Feedback Program) for adolescents and young adults with cancer. As part of this study, up to 160 adolescents and young adults (AYAs) with cancer will be randomized to one of these groups. Participants who enroll in this trial will be given an electronic pill bottle or box with a computer chip to store their medication. After using the electronic monitor for a few weeks to assess baseline adherence, participants who demonstrate non-adherence and have used the electronic monitor without difficulty will be asked to complete pre-treatment questionnaires. Next, participants will be randomly assigned to one of the two groups and complete their assigned program. Adolescents and young adults will continue to use the electronic monitor to store their medication until approximately a month after their program ends. After their program ends, participants will complete questionnaires at post-treatment and again about 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 15.00 to 24.99 years of age
* Patient is diagnosed with cancer
* Patient is prescribed an oral anticancer/antitumor agent or prophylaxis

Exclusion Criteria:

* Patient is not fluent in English
* Patient evidences significant cognitive deficits
* Patient's medical status or treatment precludes participation
* Patient enrolled on a medical trial requiring medication storage in a trial-provided container
* Patient demonstrates greater than or equal to 95% adherence during run-in period
* Patient declines to use or has difficulty using electronic adherence monitoring device during run-in

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | The 1-month period following the completion of one of the study programs.
  Each participant will be given an electronic adherence monitoring device to store their medication. An electronic adherence monitoring device is a pill bottle or box with an embedded computer chip. The computer chip records each time the device is opened. These device openings, or actuations, will be compared with the patient's prescribed medication regimen to compute their adherence (defined as the percentage of doses taken as prescribed).

SECONDARY OUTCOMES:
Quality of Life (Mental Health) | Approximately 1 month after completing one of the study programs
  PROMIS (Patient-Reported Outcomes Measurement Information System) Global Mental Health 2a. Raw score range = 2-10. Higher scores = better quality of life.
Quality of Life (Physical Health) | Approximately 1 month after completing one of the study programs
  PROMIS (Patient-Reported Outcomes Measurement Information System) Global Physical Health 2a. Raw score range = 2-10. Higher scores = better quality of life.
Healthcare Utilization | 6 months post-treatment
  Number of oncology visits, lab draws, ED visits, and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Meghan E. McGrady, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Columbia University Irving Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington